CLINICAL TRIAL: NCT01950221
Title: 12-Month, Double-blind, Placebo-Controlled Study of Pomegranate Extract
Brief Title: Pomegranate Extract and Memory
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: POM Wonderful LLC (Industry)
Responsible Party: Principal Investigator, Gary Small, MD, Professor of Psychiatry and Biobehavioral Sciences, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 11-002413; NCT01571193 (obsolete NCT alias)
Record Dates: First submitted 2013-09-16; First posted 2013-09-25 (Estimated); Last update posted 2020-03-02 (Actual); Status verified 2020-02

CONDITIONS: Healthy Volunteers
Keywords: Double-blind Trial; Placebo-controlled; Pomegranate; Memory; Memory Impairment; Cognition; Ages 50-75
MeSH Terms: conditions — Memory Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- POMx (Experimental): POMx is a 1,000 milligram capsule of natural pomegranate polyphenol extract.
  Interventions: Dietary Supplement: POMx
- Placebo (Placebo Comparator): Composition of the Drug Placebo Component/Function/Weight/Percentage of Fill Weight = Cellulose/Bulk agent/658 mg/64.5% Caramel/Colorant/79mg/7.8% Beet root/Flavor Ingredient/263mg/25.8% Magnesium stearate/USP Lubricant/10mg/1.0% Silica Dioxide/FCC Glidant/10mg/1.0% Total = 1020 mg/100% The method of manufacture of the placebo is identical to that of the drug product, except cellulose, caramel, and beet root are added in place of the active ingredient.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: POMx — "POMx" is a 1,000 milligram capsule of natural pomegranate polyphenol extract.
  Arms: POMx
Other: Placebo
  Arms: Placebo

SUMMARY:
This project is designed to study whether pomegranate extract benefits cognitive abilities in middle-aged and older non-demented volunteers. Subjects will be randomly assigned to one of two treatment groups: either a placebo or the pomegranate extract supplement. Both the placebo and pomegranate extract will be packaged in 1000 milligram capsules to maintain blindness. Subjects will take one 1000 milligram capsule daily for twelve months.

The investigators expect the people receiving the pomegranate extract supplement to show better cognitive performance compared with those receiving a placebo after one, six, and twelve months. The investigators believe cognitive decline and treatment response will vary according to a genetic risk for Alzheimer's.

The investigators will study 212 non-demented subjects aged 50-75 years. Initially, subjects will undergo a clinical assessment, an MRI and a blood draw to determine genetic risk and to rule out other neurodegenerative disorders linked to memory complaints.

Subsequently, subjects will undergo the first memory (or neuropsychological) assessments. Following the first assessment, subjects will begin taking the supplement (either the pomegranate extract or the placebo). Subjects will undergo a brief memory test at one-month mark. At six months, subjects will have a second, full neuropsychological assessment. The final assessment will take place at the end of the study, the 12-month mark. Additional blood will be drawn at baseline and at 12 months and frozen to assess inflammatory markers if outcomes are positive. Subjects will also be asked to come to the University of California, Los Angeles (UCLA) at 3 and 9 months for supplement refills.

In total, subjects will be expected to come to UCLA for 7 visits during the course of 12-13 months.

ELIGIBILITY:
Inclusion Criteria:

* Agreement to participate in the 12-month double-blind, placebo-controlled clinical trial of pomegranate extract.
* Nondemented subjects either those with normal cognition or with Mild Cognitive Impairment will be included.
* Age 50 to 75 years.
* No significant cerebrovascular disease: modified Ischemic Score of < 4
* Adequate visual and auditory acuity to allow neuropsychological testing.
* Screening laboratory tests and EKG without significant abnormalities that might interfere with the study. If screening laboratory tests or EKG show abnormalities, subject must obtain written clearance from primary care physician before continuing in the study.

Exclusion Criteria:

* Diagnosis of probable Alzheimer's disease (AD) or any other dementia (e.g., vascular, Lewy body, frontotemporal) (McKhann et al, 1984). Evidence of other neurological or physical illness that can produce cognitive deterioration. Volunteers with a history of stroke, Transient Ischemic Attack (TIA), carotid bruits, or lacunes on MRI scans will be excluded. Determination of dementia will be based on the clinical evaluation including assessment of functional abilities, and cognitive screening.
* Contraindication to the MRI including claustrophobia, metal in body, surgery within 60 days, certain implants or previous abnormal MRI results.
* Evidence of Parkinson's disease as determined by the motor examination (items 18-31) of the Unified Parkinson's Disease Rating Scale (Fahn et al, 1987).
* History of myocardial infarction within the previous year, or unstable cardiac disease.
* Uncontrolled hypertension (systolic BP > 170 or diastolic BP > 100).
* History of significant liver disease, clinically-significant pulmonary disease, or diabetes.
* Current diagnosis of any major psychiatric disorder
* Current diagnosis or history of alcoholism or substance addiction.
* Regular use of any medication that may affect cognitive functioning including: centrally active beta-blockers, narcotics, Clonidine, anti-Parkinsonian medications, antipsychotics, systemic corticosteroids, medications with significant cholinergic or anticholinergic effects, anti-convulsants, or Warfarin.
* Occasional use of anxiety or sleeping medications known to cause cognitive dulling will be allowed, but discouraged: chloral hydrate, non-benzodiazepine hypnotics such as: Ambien (Zolpidem) and Lunesta; or benzodiazepines such as Ativan (Lorazepam), Xanax (Alprazolam), Klonopin (Clonazepam), and Restoril (Temazepam).
* Use of any of the following medications: Amitriptyline, Amiodarone, Desipramine, Fenofibrate, Flecainide, Fluconazole, Fluoxetine, Fluvastatin, Fluvoxamine, Isoniazid, Lovastatin, Ondansetron, Phenylbutazone, Probenecid, Sertraline, Sulfamethoxazole, Sulfaphenazole, Teniposide, Voriconazole, Warfarin, and Zafirlukast
* Use of cognitive enhancing supplements (e.g. Ginkgo biloba).
* Use of any supplement containing pomegranate or pomegranate juice.
* Use of any investigational drugs within the previous month or longer, depending on drug half-life.
* Pregnancy.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 212 (Actual)
Dates: Start 2011-10; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Improved cognitive performance | 1 year
  Non-demented volunteers aged 50-75 who receive a daily dietary supplement of pomegranate extract will show improved cognitive performance compared to baseline versus those receiving a placebo after one, six, and twelve months.

SECONDARY OUTCOMES:
Cognitive performance improvement and genotype | 1 year
  Cognitive change in the pomegranate intervention group will vary according to genotype.

CONTACTS AND LOCATIONS:
Locations (1):
- UCLA Longevity Center, Los Angeles, California, United States

REFERENCES:
- See also: UCLA Longevity Center — http://www.semel.ucla.edu/longevity